CLINICAL TRIAL: NCT03257813
Title: Clinical Study to Evaluate the Non-inferiority of PRO-122 an Ophthlamic Solution Manufactured by Laboratorios Sophia, Previous Treatment With Krytantek Ofteno ®, in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension.
Brief Title: Non-inferiority of PRO-122 Ophthalmic Solution vs KRYTANTEK Ofteno® in Glaucoma or Ocular Hypertension (CONFORTK)
Acronym: CONFORTK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH122-0914/III
Record Dates: First submitted 2017-08-01; First posted 2017-08-22 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: timolol; dorzolamide; brimonidine; Glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Timolol; dorzolamide; Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: 60 subjects with diagnosis of open angle primary glaucoma with mild, moderate or severe damage and / or with intraocular hypertension users of Krytantek Ofteno® at least two previous months and are under control Of the corresponding IOP target.
  a study group A or B will be randomly assigned, in group A, therapy with Krytantek Ofteno® will be continued for 30 days, in which the subject will be evaluated again and switched from therapy to solution PRO-122 which will be used for 30 days until the 60th day, date of the final visit.
  In the case of those assigned to group B on day 1, the change to PRO-122 solution will be made for 30 continuous days until the date of revision on day 30, the day on which treatment with Krytantek Ofteno® will be restored to continue until the Day 60 for the final evaluation.
  The selected subjects will be observed for 60 days.
Who Masked: Participant, Investigator
Masking Description: Masking will be carried out using identical boxes in the primary package in both groups.
  Blinding for the research subject and the investigator will be carried out by using labels containing the assignation number, which will replace the original labels in the case of the comparator. Due to the nature of the primary containers of the research products, single-dose vials and multidose bottle, it is not possible to use identical labels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): In group A, therapy with Krytantek Ofteno® will be continued for 30 days, in which the subject will be retested and switched to a PRO-122 solution which will be used for 30 days until the 60th day, The final visit.
  Interventions: Drug: PRO-122; Drug: Krytantek Ofteno®
- Group B (Other): In group B, therapy with Krytantek Ofteno® will be suspended and changes for PRO-122 for 30 days, in which the subject will be retested and later switched to Krytantek Ofteno® solution which will be used for 30 days until the 60th day, The final visit.
  Interventions: Drug: PRO-122; Drug: Krytantek Ofteno®

INTERVENTIONS:
Drug: PRO-122 — 1 drop every 12 hours for 30 days of alternating treatment with 30 days
  Other Names: timolol, dorzolamide, brimonidine
Drug: Krytantek Ofteno® — 1 drop every 12 hours for 30 days of alternating treatment with 30 days
  Other Names: timolol, dorzolamide, brimonidine

SUMMARY:
Aim: To demonstrate the non-inferiority of the PRO-122 ophthalmic solution manufactured by Laboratorios Sophia S.A. de C.V. versus Krytantek Ofteno® ophthalmic solution like hypotensive therapy in subjects with primary open angle glaucoma or ocular hypertension.

Study design: a multicentric, prospective, crossover (2x2), double blind clinical study. Sample size: one hundred patients with primary open angle glaucoma or ocular hypertension. Patients in the period 1: In the first sequence 30 patients will be assigned to receive the ophthalmic solution: Krytantek Ofteno ® (timolol 0.5%%/brimonidine 0.2%/dorzolamide 2%) 1 drop B.I.D. during 30 days and the second sequence 30 patients will be assigned to receive the ophthalmic solution: PRO-122 1 drop B.I.D. during 30 days in the same period. Washout period: 20 hours. Patients in the period 2: the pharmacological intervention change to the opposite therapy for 30 days

DETAILED DESCRIPTION:
The American Academy of Ophthalmology Glaucoma Panel: The primary open angle glaucoma (POAG) is a progressive, chronic optic neuropathy in adults in which intraocular pressure (IOP) and other currently unknown factors contribute to damage and in which, in the absence of other identifiable causes, there is a characteristic acquired atrophy of the optic nerve and loss of retinal ganglion cells and their axons. This condition is associated with an anterior chamber angle that is open by gonioscopic appearance.

This is a multicentric, crossover, double blind and prospective clinical study. The investigators will include patients with confirmed diagnosis of primary open-angle glaucoma or ocular hypertension, with target intraocular pressure (TIOP) within a range at which a patient is likely to remain stable or at which worsening of glaucoma will be slow enough that the risk of additional intervention is not justified.

Patients will be randomly divided into 2 groups, one of them treated with a known formulation of timolol 0.5%/brimonidine 0.2%/dorzolamide 2% (Krytantek Ofteno®, Laboratorios Sophia, Mexico) and the other one treated with PRO-122 ophthalmic solution. Patients will receive 1 drop B.I.D. into the lower conjunctival sac of either formulations and were examined at days: 1, 15, 30, 45 and 61 after initiation of treatment. A phone call security at day 75 will be performed.

Primary efficacy outcome: To evaluate the efficacy of PRO-122 versus Krytantek Ofteno® instilled onto the ocular surface in subjects with primary open angle glaucoma (POAG) or ocular hypertension (HTO), to control and maintenance of the target intraocular pressure (TIOP).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* male or female.
* obtained in the external consultation.
* With diagnosis primary of open-angle glaucoma and / or hypertension classified as mild, moderate or severe glaucomatous damage, users of Krytantek Ofteno® at least two months prior to inclusion and under control of the target IOP.
* informed consent.

Exclusion Criteria:

General Criteria

1. Subjects with topical or systemic medication that interferes decisively in the results of the study. (Such as topical immunomodulators, lacrimal point tamponade, corticosteroids, ocular hypotensives other than those listed above, artificial tears with preservative).
2. Subjects (female) with an active sex life who are not using a contraceptive method.
3. Female Subjects in pregnancy or breastfeeding.
4. Female subjects with positive urine pregnancy test.
5. Positive drug addiction (verbal interrogation).
6. Subjects who have participated in any clinical research study in the last 40 days.
7. Legally or mentally disabled subjects to give informed consent for their participation in this study.
8. Subjects who can not comply with the appointments or with all the requirements of the protocol.

Ophthalmologic criteria

1. Subject with only one eye with vision.
2. Subjects with visual capacity 20/200 or worse.
3. Subjects with a narrow-angle history without treatment, with or without total or partial closure of the angle in either eye.
4. Subjects with corneal abnormalities that prevent applanation tonometry.
5. Subjects with ocular surgery or ocular trauma 6 months prior to inclusion.
6. Any ocular laser surgery 3 months prior.
7. Any uncontrolled or progressive retinal disease.
8. Inflammatory diseases of any kind.
9. Contact lens wearers.
10. Subjects with a history of hypersensitivity to any of the ingredients of the research product or its analogues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-06-18 (Actual)

IPD SHARING:
Plan to Share IPD: No
Confidentiality Policy

REFERENCES:
- [Derived] Gomez-Aguayo F, Paczka JA, Lenero-Cordova R, Jimenez-Roman J, Davila-Villarreal J, Hartleben C, Baiza-Duran L, Olvera-Montano O, Garcia-Velez F, Munoz-Villegas P. A Phase III Randomized Clinical Trial of a 0.5% Timolol + 0.2% Brimonidine + 2.0% Dorzolamide Fixed Combination, Preservative-Free Ophthalmic Solution vs. 0.5% Timolol + 0.2% Brimonidine + 2.0% Dorzolamide Fixed Combination in Patients with Controlled Primary Open-Angle Glaucoma. Ophthalmol Ther. 2018 Jun;7(1):145-156. doi: 10.1007/s40123-018-0128-8. Epub 2018 Apr 21. PMID 29680880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 30 | 30
Completed | 24 | 27
Not Completed | 6 | 3
Not completed — Protocol Violation | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.43 (8.86) | 64.37 (12.84) | 66.44 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  hispanic | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Intraocular pressure, Unit: Millimeters of mercury (mmHg) type of variable: Continuous, Measurement method: Goldman applanation tonometry. Normal intraocular pressure 11-21 mmHg.
  The change between the IOP of both groups was compared (sequence 1 versus sequence 2) of the data obtained at the end of each period (day 30 and day 60).
Time Frame: Change from Baseline intraocular pressure at day 30 and 60.
Population: the statistical analysis was carried out taking into account each eye as a case number, therefore, each research subject could provide 2 cases.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Groups:
- Sequence A: First Period: PRO-122: 1 drop every 12 hours for 30 days of alternating treatment with 30 days
  Second Period: Krytantek Ofteno®: 1 drop every 12 hours for 30 days of alternating treatment with 30 days
- Sequence B: First Period: Krytantek Ofteno®: 1 drop every 12 hours for 30 days of alternating treatment with 30 days
  Second Period: PRO-122: 1 drop every 12 hours for 30 days of alternating treatment with 30 days
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 48 | 54
mmHg
  basal visit (day 1) | 13.60 (2.9) | 12.13 (1.8)
  Crossover visit (day 30) | 13.19 (3.2) | 11.80 (2.1)
  Final visit (day 60) | 12.60 (3.0) | 11.24 (1.6)
Statistical Analysis 1: Comparison: Sequence A; Test type: Non-Inferiority — it will be considered not inferior if they keep the IOP goal with differences of no more than 1.5 mmHg; p = 0.013, t-test, 2 sided — Baseline
Statistical Analysis 2: Comparison: Sequence B; Test type: Non-Inferiority — it will be considered not inferior if they keep the IOP goal with differences of no more than 1.5 mmHg; p = 0.001, t-test, 2 sided — CrossOver
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — it will be considered not inferior if they keep the IOP goal with differences of no more than 1.5 mmHg; p = 0.050, t-test, 2 sided — Final Visit

2. Secondary Outcome: Visual Acuity (VA)
Description: The VA will be evaluated basally, without refractive correction with the Snellen chart. A Snellen chart is placed at a standard distance: 20 ft. At this distance, the symbols on the line representing "normal" acuity subtend. This line, designated 20/20 is the smallest line that a person with normal acuity can read at a distance of 20fs. the scale consists of 11 lines of letters of different size, the size of the letter gives a fractional value according to the visual acuity of the patient, the value is inversely proportional to the visual acuity, if the denominator is greater the visual acuity will be less.
  Line 1: 20/200 Line 2: 20/100, Line 3: 20/70, line 4: 20/50, line 5: 20/40, Line 6: 20/30, line 7: 20/25, Line 8: 20/20, line 9: 20/15, line 10: 20/13, line 11: 20/10. the differences between groups in the basal, cross over and final visit will be evaluated.
Time Frame: Visual Acuity at Baseline (day 1) crossover visit (day 30) and final visit (day 60)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: eyes
Groups:
- Sequence B: First Period: Krytantek Ofteno®: 1 drop every 12 hours for 30 days of alternating treatment with 30 days
  Second Period: _1 drop every 12 hours for 30 days of alternating treatment with 30 days
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 48 | 54
score on a scale
  basal visit (day 1) | 38.31 (3.577) | 39.48 (3.742)
  Crossover visit (day 30) | 36.85 (3.806) | 40.43 (3.753)
  Final visit (day 60) | 38.98 (3.717) | 35.50 (3.402)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — to be considered as not inferior to the group, the differences between both should not be greater than 2 points on the snellen scale; p = 0.823, t-test, 2 sided — Baseline
Statistical Analysis 2: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.507, t-test, 2 sided — CrossOver
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.495, t-test, 2 sided — Final Visit

3. Other Pre Specified Outcome: Adverse Events
Description: The presence of adverse events by percentage between groups will be evaluated. the scale is present or absent.
Time Frame: 75 days, includes the security call
Population: the statistical analysis was carried out taking into account each eye as a case number, therefore, each research subject could provide 2 cases. statistical analysis by intention to treat (ITT)
Measure: Number; unit: percentage of adverse events
Units Other Than Participants: eyes
Groups:
- PRO-122: all subjects who received at least one application of PRO-122 in both sequences
- Krytantek Ofteno: all subjects who received at least one application of Krytantek Ofteno in both sequences
Arm/Group | PRO-122 | Krytantek Ofteno
Number analyzed (Participants) | 60 | 60
Number analyzed (eyes) | 120 | 120
percentage of adverse events
  mild | 55.6 | 18.2
  moderate | 44.4 | 72.7
  severe | 0 | 9.1
Statistical Analysis 1: Comparison: PRO-122 vs Krytantek Ofteno; Test type: Non-Inferiority — to be considered as not inferior to the group, the differences between both should not be greater than 20% of the frequency; p = 0.085, Chi-squared

4. Other Pre Specified Outcome: Conjunctival Hyperemia
Description: the conjunctival hyperemia will be evaluated by the presence or absence of it and the percentage of affected by group will be reported.
Time Frame: Baseline (day 1) crossover visit (day 30) and final visit (day 60)
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 49 | 60
percentage of eyes
  basal visit (day 1) | 39.6 | 11.1
  Crossover visit (day 30) | 37.5 | 25.9
  Final visit (day 60) | 20.8 | 13.0
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.001, Fisher Exact — Baseline
Statistical Analysis 2: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.148, Fisher Exact — CrossOver
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.212, Fisher Exact — Final Visit

5. Other Pre Specified Outcome: Chemosis
Description: Chemosis: qualitative ordinal variable, will be evaluated by the presence or absence of it and the percentage of affected by group will be reported.
Time Frame: Baseline (day 1) crossover visit (day 30) and final visit (day 60)
Population: as for outcome 1
Measure: Number; unit: percentage of chemosis
Units Other Than Participants: eyes
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 49 | 50
percentage of chemosis
  basal visit (day 1) | 0 | 3.7
  Crossover visit (day 30) | 0 | 3.7
  Final visit (day 60) | 0 | 0
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.497, Chi-squared, Corrected — Baseline
Statistical Analysis 2: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.497, Chi-squared, Corrected — CrossOver
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0, Chi-squared, Corrected — Final Visit No statistic will be calculated because Final Chemosis is a constant

6. Other Pre Specified Outcome: Eye Burning
Description: Eye ocular burning will be evaluated by the presence or absence of it and the number of affected by group will be reported.
Time Frame: Baseline (day 1) crossover visit (day 30) and final visit (day 60)
Population: as for outcome 1
Measure: Number; unit: number of eye burning
Units Other Than Participants: eyes
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 49 | 50
number of eye burning
  basal visit (day 1) | 16 | 18
  Crossover visit (day 30) | 12 | 18
  Final visit (day 60) | 14 | 19
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 1.000, Chi-squared — baseline
Statistical Analysis 2: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.391, Chi-squared — Cross Over
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.534, Chi-squared — Final Visit

7. Other Pre Specified Outcome: Number of Eyes With Tearing
Description: Tearing will be evaluated by the presence or absence of it and the number of affected by group will be reported
Time Frame: Baseline (day 1) crossover visit (day 30) and final visit (day 60)
Population: as for outcome 1
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 49 | 50
eyes
  basal visit (day 1) | 9 | 2
  Crossover visit (day 30) | 8 | 9
  Final visit (day 60) | 7 | 9
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.023, Chi-squared, Corrected — Baseline
Statistical Analysis 2: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 1.000, Chi-squared — CrossOver
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.793, Chi-squared — Final Visit

8. Other Pre Specified Outcome: Number of Eyes With Foreign Body Sensation
Description: Foreign body sensation will be evaluated by the presence or absence of it and the number of affected by group will be reported.
Time Frame: Baseline (day 1) crossover visit (day 30) and final visit (day 60)
Population: as for outcome 1
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 49 | 50
eyes
  basal visit (day 1) | 14 | 14
  Crossover visit (day 30) | 14 | 16
  Final visit (day 60) | 5 | 7
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.825, Chi-squared — Baseline
Statistical Analysis 2: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 1.000, Chi-squared — CrossOver
Statistical Analysis 3: Comparison: Sequence A vs Sequence B; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.765, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 months
Description: The study's e-CRF was designed to collect adverse events for each research product separately. The sequence or crossing of the products under investigation was not considered for the report of adverse events because it can be detected at what time the event occurs and directly link it to the product that was being administered at the same time.
Groups:
- PRO-122: All adverse events that occurred with the product under investigation PRO-122 were collected regardless of the sequence in which they participated.
  The 30 participants of both sequences received at least one dose of PRO-122, therefore 60 subjects exposed in this group are considered.
- Krytantek Ofteno®: All adverse events that occurred with the product under investigation Krytantek Ofteno® were collected regardless of the sequence in which they participated.
  The 30 participants of both sequences received at least one dose of Krytantek Ofteno®, therefore 60 subjects exposed in this group are considered.
Arm/Group | PRO-122 | Krytantek Ofteno®
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/60
Other Adverse Events (participants affected / at risk) | 12/60 | 8/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-122 (N=60) | Krytantek Ofteno® (N=60)
acute gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — presented with acute abdominal pain, was hospitalized with a presumptive diagnosis of appendicitis; appendicitis is ruled out and the diagnosis of acute gastritis is given, receiving treatment and resolved without sequelae.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-122 (N=60) | Krytantek Ofteno® (N=60)
headache (General disorders) | 2 (2) | 0 (0)
Meniere syndrome exacerbated (General disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
atopic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rhinopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
allergic Blepharokeratoconjunctivitis (Eye disorders) | 2 (2) | 0 (0)
pharyngitis tonsillitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
maxillary traumatism (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bacterial conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dotted Keratopathy (Eye disorders) | 0 (0) | 3 (3)
stomach flu (Gastrointestinal disorders) | 1 (1) | 0 (0)
atopic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
intestinal amebiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
peptic acid disease (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03257813/Prot_SAP_000.pdf